CLINICAL TRIAL: NCT04744805
Title: Mask-associated Dry Eye Symptoms: an Online Survey of 6262 Chinese Persons
Brief Title: Mask-associated Dry Eye Symptoms in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021003
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Masks; Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mask wear
  Interventions: Other: face mask or not
- dry eye
  Interventions: Other: face mask or not

INTERVENTIONS:
Other: face mask or not — long term face mask wear

SUMMARY:
To review the relationship of increased face mask usage arising from lockdown measures instituted during the COVID-19 pandemic with dry eye symptoms on Chinese people, and make recommendations for mitigating potential detrimental effects on dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age >=8 years mental health

Exclusion Criteria:

* eye diseases mental or systemic diseases

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An online survey of persons focused on face mask usage
Sampling Method: Probability Sample
Enrollment: 6262 (Estimated)
Dates: Start 2021-01-29 (Estimated); Primary Completion 2021-02-05 (Estimated); Study Completion 2021-02-06 (Estimated)

PRIMARY OUTCOMES:
time of face mask wear | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Director — Tianjin Eye Hospital

REFERENCES:
- [Derived] Fan Q, Liang M, Kong W, Zhang W, Wang H, Chu J, Fang X, Song Y, Gao W, Wang Y. Wearing face masks and possibility for dry eye during the COVID-19 pandemic. Sci Rep. 2022 Apr 13;12(1):6214. doi: 10.1038/s41598-022-07724-0. PMID 35418586